CLINICAL TRIAL: NCT02863224
Title: Advanced Glycation End Products as a Biomarker for Accelerated Ageing in Glaucomatous Optic Neuropathy
Brief Title: Advanced Glycation End Products as a Biomarker for Accelerated Ageing
Status: Completed | Type: Observational
Sponsor: University of Plymouth (Other)
Responsible Party: Principal Investigator, Leanne Smewing, Principal Investigator, University of Plymouth
Other Study IDs: 204642
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Primary Open Angle Glaucoma; Normal Tension Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Low Tension Glaucoma; Ocular Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples will be analysed within the study time frame. They will be used for this study only and will be destroyed as per HTA guidelines once no longer needed for this study.

GROUPS / COHORTS (4):
- Healthy control
- Ocular hypertension
- Primary open angle glaucoma
- Normal tension glaucoma

SUMMARY:
Globally primary open angle glaucoma (POAG) affects over 60 million people. The exact pathogenesis of POAG is poorly understood. A significant risk factor for glaucoma is advancing age. The rate of ageing is not the same in all age matched individuals. The concept of accelerated ageing suggests that the presence of a number of specific genetic, environmental or systemic risk factors may cumulate to accelerate the ageing process in some individuals and lead to the development of age-related disease. Understanding the factors that influence accelerated ageing is vital.

Advanced glycation end products (AGEs) are a complex group of compounds that are naturally formed. They accumulate gradually with age in cells, tissues and blood vessels throughout the body where they adversely affect structure and function. Circulating AGE levels can be influenced by oxidative stress levels and dietary intake. Recent research has found that sustained exposure to high levels of circulating AGEs could be a major factor in the development of a number of chronic age-related degenerative disorders, including POAG.

To date there have been few clinical studies that have been able to non-invasively explore the association between AGE levels and the development and progression of glaucomatous optic neuropathy (GON), or to explore the possible contribution that oxidative stress and dietary intake make to total tissue AGE levels in such patients. Furthermore little is understood about the relationship between AGE levels and retinal vascular function, a parameter known to be altered in GON that also could be influenced by AGE levels.

The proposed study will aim to evaluate whether tissue-bound AGE levels are associated with parameters of retinal vascular function, oxidative stress, dietary intake and the presence of GON. Establishing this association could increase our understanding of the pathogenesis of GON and allow a new biomarker for accelerated ocular ageing to be realised

ELIGIBILITY:
Inclusion Criteria:

* Must have had an eye test within the last two years
* Aged 50+
* Informed, written consent
* Have adequate understanding of English language to be able to comprehend the oral and written instructions.
* Participants must be able to complete a 12-hour overnight fast, which includes no alcohol or caffeine.

Inclusion criteria for Ocular hypertension, Primary open angle glaucoma and normal tension glaucoma:

- Follows guidelines set out within the protocol and used at Derriford REI

Exclusion Criteria:

* Diabetes
* Current smokers
* History of stroke/TIA
* Coronary artery disease/heart failure/arrhythmia/angina
* Peripheral vascular disease
* Severe dyslipidaemia
* Hyper/hypothyroidism

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy controls, ocular hypertension, primary open angle glaucoma and normal tension glaucoma groups aged 50 years and older will be studied. Different parameters will be looked at with an aim to understand ageing in glaucomatous optic neuropathy.
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Tissue bound AGE level (AU) | Tissue bound AGE level (AU) will be measured for each participant at their second session (within 3 months of volunteering).
  Level of AGE found in the skin - measured from the lower portion of the arm

CONTACTS AND LOCATIONS:
Locations (1):
- Plymouth University, Plymouth, Devon, United Kingdom